CLINICAL TRIAL: NCT01711008
Title: The Effect of Breakfast Size Prior to Morning Exercise on Cognition, Mood and Appetite Later in the Day in Habitually Active Women
Brief Title: The Effect of Breakfast Size Prior to Morning Exercise on Cognition, Mood and Appetite in Habitually Active Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Rachel Veasey, MSc, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 29W5
Record Dates: First submitted 2012-09-25; First posted 2012-10-19 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Alteration of Cognitive Function
Keywords: Breakfast size; Exercise; Cognitive performance; Mood; Appetite; Active women
MeSH Terms: conditions — Motor Activity | interventions — Edible Grain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Breakfast (Placebo Comparator): Water only
  Interventions: Dietary Supplement: No breakfast
- 20g Cereal (Active Comparator): 20g Kelloggs Special K cereal with 83ml semi-skimmed milk
  Interventions: Dietary Supplement: Cereal
- 40g Cereal (Active Comparator): 40g Kelloggs Special K cereal with 166ml semi-skimmed milk
  Interventions: Dietary Supplement: Cereal

INTERVENTIONS:
Dietary Supplement: Cereal
  Other Names: Breakfast cereal
  Arms: 20g Cereal; 40g Cereal
Dietary Supplement: No breakfast
  Arms: No Breakfast

SUMMARY:
Both regular exercise and breakfast consumption have well known health benefits. Consuming breakfast prior to morning exercise may influence appetite, mood and cognitive function later in the day. The purpose of this study is to test whether the amount of food consumed at breakfast prior to exercise influences these parameters in active women.

ELIGIBILITY:
Inclusion Criteria:

* Must be habitually active (exercising for least 30 minutes, 3 times per week for at least the previous 6 months)
* Must have a normal exercise routine includes a minimum of 1 morning exercise session (which takes place between 6am-11am) each week
* Must run on a regular basis (at least once per week) and be able to run at a moderate pace for 30 minutes non-stop on a treadmill
* Must consume breakfast on most days of the week, usually consume breakfast before undertaking a morning exercise session and be comfortable consuming a bowl of cereal 45mins before running

Exclusion Criteria:

* English not first language
* Smoking
* Previous or current eating disorders, metabolic disorders, gastric problems or any contraindications of exercise.
* Pregnancy
* The habitual use of some prescription or over the counter medications (excluding contraception) or herbal/dietary supplements (please ask the researcher)
* A history of or current learning difficulties, ADHD or dyslexia
* Daily use of an inhaler to control asthma
* Allergies or intolerances to any of the foods provided in the study (Special K cereal, semi-skimmed milk, pasta, tomato sauce, cheese, olive oil, rice, custard)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive function change from baseline scores | Assessed hourly until 4.5 hours and at 6.5 and 10.5 hours
  Participants will complete 4 cognitive tasks (Four Choice Reaction Time, NBack, Stroop and RVIP) measuring reaction time, short-term memory, speed of processing and attention.

SECONDARY OUTCOMES:
Mood change from baseline scores | Assessed hourly until 4.5 hours and at 6.5 and 10.5 hours
  Mood will be assessed using Visual Analogue Scales (VAS) immediately before and after each set of cognitive tasks.

OTHER OUTCOMES:
Appetite change from baseline scores | Assessed hourly until 4.5 hours and at 6.5 and 10.5 hours
  Appetite will be assessed using Visual Analogue Scales (VAS) immediately before each set of cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Veasey, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria Univerity, Newcastle upon Tyne, Tyne and Wear, United Kingdom